CLINICAL TRIAL: NCT01405573
Title: Sorafenib in the First Line Treatment of Advanced Hepatocellular Carcinoma With Child-Pugh Liver Function Class B: Multicentre Phase 3 Randomized Trial
Brief Title: Sorafenib in First-line Treatment of Advanced B Child Hepatocellular Carcinoma
Acronym: BOOST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of enrolment
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOOST; EudraCT number 2009-013870-42 (Registry Identifier: EudraCT)
Record Dates: First submitted 2010-02-26; First posted 2011-07-29 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Advanced Adult Hepatocellular Carcinoma
Keywords: Child Pugh B; first line
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Best Supportive Care (Active Comparator): best supportive care
  Interventions: Other: Best Supportive Care
- B: Sorafenib 400 mg, twice a day + Best Supportive Care (Experimental): sorafenib + best supportive care
  Interventions: Other: Best Supportive Care; Drug: sorafenib

INTERVENTIONS:
Other: Best Supportive Care — Therapy given according to clinical practices at participating centres. Experimental therapies not permitted.
Drug: sorafenib — 400 mg twice a day
  Arms: B: Sorafenib 400 mg, twice a day + Best Supportive Care

SUMMARY:
The purpose of this study is to to compare the addition of sorafenib (800 mg/day)to best supportive care with best supportive care alone in terms of survival in patients with hepatocellular carcinoma (HCC) with impaired liver function (Child B).

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third cause of death for cancer in the world with an increasing incidence. No systemic therapy has proven effective in patients with advanced HCC until 2007, when results of the SHARP trial were presented. In this trial, the orally active multi-kinase inhibitor sorafenib (800 mg/day) significantly prolonged survival compared with placebo in patients with advanced HCC and good liver function (Child A). The same authors concluded that the effect of the drug in the population of patients with more impaired liver function should be further studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of hepatic cell carcinoma (HCC) according to the AASLD- EASL criteria
* Age >18 years
* Advanced stage of disease defined as HCC not eligible for locoregional treatments (ab initio or following progression after such treatments)
* Liver function classified as Child-Pugh class B
* ECOG performance status < or = 2
* Life expectancy of at least 2 months
* Adequate contraception for fertile male and female patients
* Signed informed consent

Exclusion Criteria:

* Prior exposure to sorafenib or antiangiogenesis drugs
* Concomitant diseases that contraindicate the use of sorafenib
* Gastro-intestinal bleeding in the previous 30 days
* Altered renal function(creatinine > 1.5 x ULN), or haematological function (platelet count < 60 x 10^9/L, hemoglobin < 9 g/dl)
* Serious active infections (> grade 2 CTCAE version 3.0)
* Congestive heart failure, history of congestive heart failure, unstable angina pectoris, myocardial infarct or significant valvular heart disease or uncontrolled heart arrhythmia
* Patients who are unable or unwilling to participate in the study
* Pregnant or lactating females
* Hepatic encephalopathy of any grade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
overall survival | 6 months

SECONDARY OUTCOMES:
worst grade toxicity per patient | every 4 weeks
  worst grade toxicity (according to Common Terminology Criteria for Adverse Events version 4.03) per patient in both treatment arms
quality of life | every 4 weeks for 6 months
progression free survival | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Daniele, M.D., Principal Investigator — Azienda Sanitaria Rummo, Benevento, Division of Medical Oncology; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D, Principal Investigator — Second University of Naples, Italy; Chair of Medical Statistics; Antonio Gasbarrini, M.D., Principal Investigator — Università Cattolica del S. Cuore, Policlinico Gemelli, Roma; Giacomo Carteni', M.D., Principal Investigator — Ospedale Antonio Cardarelli, Napoli
Locations (25):
- Italy (25):
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Policlinico Giaccone, Palermo, PA
  - S. Orsola-Malpighi, Bologna
  - Ospedale Ramazzini di Carpi, Carpi
  - Osp. Civile Infermi, Faenza
  - Azienda Ospedaliera Careggi, Florence
  - IRCCS-Azienda Ospedaliera Universitaria San Martino-IST, Genova
  - AO C. Poma, Mantova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - A.O.U. G.Martino- Policlinico Universita di Messina, Messina
  - Istituto Nazionale Tumori, Milan
  - A.O.U. Federico II, Napoli
  - AOU II Università di Napoli, Napoli
  - Istituto Nazionale dei Tumori, Napoli
  - Ospedale Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Istituto Oncologico Veneto, Padua
  - A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale Guglielmo da Saliceto, Piacenza
  - AO S. Carlo, Potenza
  - Policlinico Universitario Tor Vergata, Roma
  - Oncologia IRCCS - Casa Sollilevo Sofferenza, S. Giovanni Rotondo
  - Azienda Ospedaliera Universitaria Arcispedal, U.O. di Oncologia Clinica, Sant'Anna Di Ferrara
  - A.O. Trevigilio - Caravaggio, Trevigilio